CLINICAL TRIAL: NCT00057512
Title: Open-Label Phase 1 Dose Escalation Study of Intralesional Injection of M4N in Patients With Refractory Malignant Tumors of the Head and Neck
Brief Title: Study of Intralesional Injection of M4N in Patients With Refractory Malignant Tumors of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erimos Pharmaceuticals (Industry)
Collaborators: Duke University (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M4N001
Record Dates: First submitted 2003-04-03; First posted 2003-04-04 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2006-01

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — terameprocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intratumoral M4N (Experimental): The initial dose was 5 mg/cm3 of tumor volume on Days 1, 8, and 15. Dose escalation in cohorts on this schedule took place up to 20 mg/cm3 tumor volume. The dose per lesion was based upon the volume of tumor, and the total dose did not exceed 1197 mg M4N/m2 body surface area.
  Interventions: Drug: M4N

INTERVENTIONS:
Drug: M4N — Dose escalation study of M4N administered intratumorally on days 1, 8 and 15. Dose escalated in cohorts on three weeks schedule to a target of 20 mg/cm3 tumor volume.
  Other Names: Tetra-O-Methyl Nordihydroguaiaretic Acid or EM-1421

SUMMARY:
The purpose of this study will be to determine the safety and tolerability of intratumoral M4N. Patients suffering from cancer of the head and neck that is recurrent after primary treatment with surgery, radiation therapy, and/or chemotherapy may be eligible. The design is a Phase 1 dose escalation study of M4N administered intratumorally once weekly, initially for three weeks. Dose will be escalated on the starting schedule to a target of 20 mg/cm3 tumor volume and then, new patient cohorts will have their schedule extended to weekly M4N for 4 weeks. Dose escalation will continue, assuming tolerability, so that cohorts will be treated for 6 weeks, and finally, 8 weeks.

DETAILED DESCRIPTION:
Study data collected will include pre-study demographics and measurements, treatment compliance, efficacy determined by tumor measurements, M4N levels in blood for pharmacokinetics, serum and biochemical determinations, hematology determinations, and patient vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age.
* Patients with documented histologic evidence of head and neck cancer with clinically measurable disease. Head and neck cancer could have been recurrent after primary treatment with surgery, radiation therapy and/or chemotherapy.
* Measurable tumor by direct inspection, photography, or by imaging (CT scan or MRI).
* Life expectancy of at least 3 months in the Investigators' opinion.
* Negative pregnancy test if in women of childbearing potential within 1 week of starting therapy.
* Patients had provided written informed consent to participate in study.
* ECOG Performance Status of 0, 1, or 2.
* Absolute neutrophil ≥ 1500/uL, hemoglobin ≥ 8 gm%, platelets ≥ 50,000/uL,
* ALT/AST ≤ 3 x ULN (upper limit of the normal range), bilirubin ≤ 1.5 x ULN and creatinine ≤ 1.5 x ULN, PT and PTT within normal limits.

Exclusion Criteria:

* Women who were pregnant or nursing.
* Women of child bearing potential who were unwilling to use an adequate method of contraception during the course of the study.
* Treatment with prior investigational agent within 30 days of entering the study.
* Patients who are unable to comply with the study requirements.
* Patients with known sensitivity to any of the study medication components.
* Patients not consenting to photography.
* Patients with tumors that have enveloped the carotid artery or whose anatomy had been distorted such that in the Investigator's opinion present high-risk of perforation or compromise during injection.
* Prior chemotherapy, radiation therapy, or surgery for the primary carcinoma within 30 days of dosing and/or had not recovered from prior therapy toxicities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MUSC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No